CLINICAL TRIAL: NCT01858935
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Escalating Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ND-L02-s0201 Injection, a Vitamin A-Coupled Lipid Nanoparticle Containing siRNA Against HSP47, in Healthy Normal Subjects
Brief Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Escalating Single Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ND-L02-s0201 Injection in Normal Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nitto Denko Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: ND-L02-s0201-001
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- ND-L02-s0201 Injection 0.03 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.1 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.2 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.4 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.5 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.6 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- ND-L02-s0201 Injection 0.8 mg/kg (Experimental)
  Interventions: Drug: ND-L02-s0201 Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ND-L02-s0201 Injection — Single IV infusion.
  Other Names: BMS-986263
  Arms: ND-L02-s0201 Injection 0.03 mg/kg; ND-L02-s0201 Injection 0.1 mg/kg; ND-L02-s0201 Injection 0.2 mg/kg; ND-L02-s0201 Injection 0.4 mg/kg; ND-L02-s0201 Injection 0.5 mg/kg; ND-L02-s0201 Injection 0.6 mg/kg; ND-L02-s0201 Injection 0.8 mg/kg
Drug: Placebo — Single IV infusion.
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety, tolerability, and pharmacokinetics of ND-L02-s0201 in normal, healthy, subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged between 18 and 55 years.
2. Willing and able to comply with the study procedures and visit schedule, including follow-up visits.
3. Able to communicate effectively with the study site personnel.
4. Body mass index (BMI) within the range of ≥18.5 and ≤30.
5. Determined by the Investigator to be in good health as documented by the following:

   1. Medical history;
   2. Physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems);
   3. Vital sign assessments: systolic blood pressure ≤140 mmHg, diastolic blood pressure ≤90 mmHg, heart rate 45-85 bpm;
   4. Normal 12-lead electrocardiogram (ECG): heart rate: 44-85 bpm, PR interval: ≤210 msec, QRS duration: ≤120 msec, QTcF: ≤430 msec;
   5. Clinical laboratory assessments within the laboratory's limits of normal values or not considered clinically significant by the Investigator; and
   6. By general observations. For any abnormalities or deviations outside the normal ranges for any clinical tests (including all laboratory tests, ECG, vital signs), the test may be repeated at the discretion of the Investigator, but the results must be discussed with the Sponsor's Medical Monitor before being judged to be not clinically significant for study participation.
6. Serum calcium, parathyroid hormone, testosterone within the laboratory's limits of normal values and 25OH-vitamin D ≥18 ng/mL.
7. Non-smoker, defined as no smoking within the 3 months prior to administration of study drug and urine cotinine < 400 ng/mL.
8. Consumed an average of no more than 2 drinks per day within the 6 months prior to administration of study drug. A drink is one 12 oz. beer, 4 oz. of wine, 1.5 oz. of 80-proof spirits, or 1 oz. of 100-proof spirits.
9. Subjects with female partners of childbearing potential must agree to use an effective barrier method of contraception (e.g., condom with spermicide) from study drug administration until the Day 28 visit. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
10. Subjects must give written informed consent.

Exclusion Criteria:

1. Any disease or condition (medical or surgical) which, in the opinion of the Investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of ND-L02-s0201, or would place the subject at increased risk.
2. History of bone disease, including osteoporosis and osteomalacia, Paget's disease of bone, or a history of unexplained fractures or fractures after minimal trauma.
3. The presence of abnormal laboratory values considered to be clinically significant by the Investigator.
4. Positive screen for Hepatitis B (HBsAg, Hepatitis B Surface Antigen), Hepatitis C (anti-HCV, Hepatitis C Antibody) or human immunodeficiency virus (HIV) (anti-HIV 1/2).
5. Participating in a concurrent interventional study with the last intervention occurring within 30 days prior to administration of study drug.
6. Received any drug therapy (including prescription and over-the-counter drugs and herbal supplements) within 1 week or 5 half-lives (whichever is longer), prior to administration of study drug. Use of non-steroidal anti-inflammatory drugs (NSAIDs), sulfonamides, probenecid or other drugs known to alter renal or tubular function is specifically prohibited for at least 5 half-lives prior to the administration of study drug. Use of immuno-suppressants is specifically prohibited within 1 week or 5 half-lives (whichever is longer), prior to administration of study drug. Vitamin A containing multi-vitamins must be withheld from Day -1 through Day 5.
7. Consumption of alcohol within 48 hours prior to administration of study drug or during the in-patient period.
8. Positive urine screen for drugs of abuse, to include ethanol, cocaine, tetrahydrocannabinol (THC), barbiturates, amphetamines, benzodiazepines, opiates, cotinine, and other drugs of abuse in the study site's location.
9. History, within the last 2 years, of alcohol abuse, significant mental illness, or physical dependence on any opioid.
10. Illicit drug use within the last 90 days.
11. Demonstration, in the opinion of study staff, of veins unsuitable for repeated venipuncture or intravenous infusion (e.g., veins that are difficult to locate, access or puncture; veins with a tendency to rupture during or after puncture).
12. Recent treatment with alternative therapies, which, in the opinion of the Investigator, could potentially confound clinical or laboratory assessments.
13. Donation or loss of more than 500 mL of blood within 56 days prior to administration of study drug or donation of plasma within 7 days prior to administration of study drug.
14. History of malignancy within the last 5 years, with the exception of non-facial basal cell carcinoma.
15. History of severe allergic or anaphylactic reactions.
16. Any other reason that, in the opinion of the Investigator or the Sponsor's Medical Monitor, makes the subject unsuitable for enrollment.
17. History of hypersensitivity to H2-receptor antagonists.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events and abnormal clinical laboratory tests | After single-ascending doses

SECONDARY OUTCOMES:
Pharmacokinetic profile and parameters | After single-ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles Phase One Services, LLC
Locations (1):
- Quintiles Phase One Services, LLC, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No